CLINICAL TRIAL: NCT05337137
Title: A Phase 1/2, Safety Confirmation, Placebo-controlled, Randomized Study of Nivolumab in Combination With Relatlimab and Bevacizumab in Treatment-naive Advanced/Metastatic Hepatocellular Carcinoma
Brief Title: A Study of Nivolumab and Relatlimab in Combination With Bevacizumab in Advanced Liver Cancer
Acronym: RELATIVITY-106
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA224-106; 2021-003606-53 (EudraCT Number); U1111-1267-1579 (Other: WHO)
Expanded Access: NCT05170659 (No longer available)
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; HCC; Liver Cancer; Relatlimab; Nivolumab; Bevacizumab; First line HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — relatlimab; Nivolumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Relatlimab + Nivolumab + Bevacizumab (Experimental)
  Interventions: Drug: Relatlimab; Drug: Nivolumab; Drug: Bevacizumab
- Arm B: Placebo + Nivolumab + Bevacizumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Bevacizumab; Other: Placebo

INTERVENTIONS:
Drug: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
  Arms: Arm A: Relatlimab + Nivolumab + Bevacizumab
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Drug: Bevacizumab — Specified dose on specified days
  Other Names: Avastin
Other: Placebo — Specified dose on specified days
  Arms: Arm B: Placebo + Nivolumab + Bevacizumab

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of triplet therapy of nivolumab, relatlimab and bevacizumab versus nivolumab and bevacizumab in participants with untreated advanced/metastatic hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced/metastatic hepatocellular carcinoma (HCC)
* Naïve to systemic therapy for advanced/metastatic HCC (prior neo-adjuvant or adjuvant immunotherapy is permitted if recurrence occurs ≥ 6 months after treatment completion and the case is discussed with BMS medical team)
* Child-Pugh score of 5 or 6 (ie, Child-Pugh A)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC
* Prior allogenic stem cell or solid organ transplantation
* Untreated symptomatic central nervous system (CNS) metastases
* Clinically significant ascites as defined by:

  i) Prior ascites that required treatment and requires on-going prophylaxis, or ii) Current ascites requiring treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 6 weeks
Overall Response Rate (ORR) by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Assessed up to 3 years

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by BICR per RECIST v1.1 in all randomized participants that are lymphocyte activation gene 3 (LAG-3) positive | Assessed up to 3 years
PFS by BICR per RECIST v1.1 in all randomized participants | Assessed up to 3 years
ORR by BICR per RECIST v1.1 in all randomized participants that are LAG-3 positive | Assessed up to 3 years
Overall Survival (OS) of all randomized participants | Assessed up to 3 years
OS of all randomized participants that are LAG-3 positive | Assessed up to 3 years
Number of participants with adverse events (AEs) | Up to 135 days after participant's last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (61):
- United States (10):
  - Local Institution - 0042, Los Angeles, California
  - Local Institution - 0039, Los Angeles, California
  - Local Institution - 0034, San Francisco, California
  - Local Institution - 0030, Washington D.C., District of Columbia
  - Local Institution - 0059, Baltimore, Maryland
  - Local Institution - 0060, Boston, Massachusetts
  - Local Institution - 0065, Boston, Massachusetts
  - Local Institution - 0061, New York, New York
  - Local Institution - 0062, The Bronx, New York
  - Local Institution - 0033, Milwaukee, Wisconsin
- Australia (5):
  - Local Institution - 0045, Camperdown, New South Wales
  - Local Institution - 0022, Adelaide, South Australia
  - Local Institution - 0026, Heidelberg, Victoria
  - Local Institution - 0013, Melbourne, Victoria
  - Local Institution - 0017, Nedlands, Western Australia
- Canada (2):
  - Local Institution - 0025, Edmonton, Alberta
  - Local Institution - 0009, Toronto, Ontario
- China (2):
  - Local Institution - 0064, Guangzhou, Guangdong
  - Local Institution - 0066, Xi'an, Shan3xi
- France (6):
  - Local Institution - 0021, Avignon, Cedex 9
  - Local Institution - 0012, Grenoble
  - Local Institution - 0001, Nice
  - Local Institution - 0002, Reims
  - Local Institution - 0008, Rennes
  - Local Institution - 0054, Suresnes
- Germany (4):
  - Local Institution - 0051, Düsseldorf, North Rhine-Westphalia
  - Local Institution - 0035, Frankfurt
  - Local Institution - 0057, Mainz
  - Local Institution - 0055, Munich
- Hong Kong (2):
  - Local Institution - 0004, Hong Kong
  - Local Institution - 0031, Shatin
- Italy (3):
  - Local Institution - 0036, Milan
  - Local Institution - 0003, Padua
  - Local Institution - 0010, Roma
- Japan (6):
  - Local Institution - 0047, Kashiwa-shi, Chiba
  - Local Institution - 0048, Matsuyama, Ehime
  - Local Institution - 0058, Kanazawa, Ishikawa-ken
  - Local Institution - 0050, Yokohama, Kanagawa
  - Local Institution - 0041, Sayama, Osaka
  - Local Institution - 0063, Chuo-ku, Tokyo
- Poland (3):
  - Local Institution - 0028, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0016, Warsaw, Masovian Voivodeship
  - Local Institution - 0023, Gdansk
- Puerto Rico (2):
  - Local Institution - 0052, Rio Piedras, PR
  - Local Institution - 0019, San Juan
- Singapore (4):
  - Local Institution - 0029, Singapore
  - Local Institution - 0027, Singapore
  - Local Institution - 0018, Singapore
  - Local Institution - 0044, Singapore
- South Korea (2):
  - Local Institution - 0037, Seongnam-si, Gyeonggido
  - Local Institution - 0056, Seoul
- Spain (6):
  - Local Institution - 0032, Santiago de Compostela, A Coruña
  - Local Institution - 0007, Santander, Cantabria
  - Local Institution - 0067, Madrid, Sede Madrid
  - Local Institution - 0053, Madrid
  - Local Institution - 0038, Pamplona
  - Local Institution - 0040, Zaragoza
- Taiwan (4):
  - Local Institution - 0043, District Taichung City, Tai Zhong Shi
  - Local Institution - 0024, Taichung
  - Local Institution - 0046, Taipei
  - Local Institution - 0049, Taipei

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com